CLINICAL TRIAL: NCT03435094
Title: A Non-interventional Two-arm Two-centre, Retrospective/Prospective Study to Compare the Effect of Alendronate 70mg Formulation (Tablet vs Effervescent Tablet) on Bone Turnover Markers and Patient Reported Outcomes
Brief Title: Effect of Alendronate 70mg Formulation on Bone Turnover Markers and Patient Reported Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Labatec Pharma SA (Industry)
Responsible Party: Sponsor
Other Study IDs: LAB-BIN-001
Record Dates: First submitted 2018-02-01; First posted 2018-02-15 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Alendronate; Tablets

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fosamax®: 1 group will be treated with alendronate 70 mg tablets (Fosamax®)
  Interventions: Drug: Fosamax 70Mg Tablet
- Binosto®: 1 group will be treated with alendronate 70 mg effervescent tablets for buffered solution (Binosto®)
  Interventions: Drug: Binosto 70Mg Effervescent Tablet

INTERVENTIONS:
Drug: Binosto 70Mg Effervescent Tablet — Assess the effect of alendronate 70mg effervescent tablet on bone turnover markers and patient reported outcomes.
  Groups: Binosto®
Drug: Fosamax 70Mg Tablet — Assess the effect of alendronate 70mg tablet on bone turnover markers and patient reported outcomes.
  Groups: Fosamax®

SUMMARY:
Compare the data obtained with two formulations of alendronate 70 mg (tablets vs effervescent tablet for buffered solution) on the change in bone turnover markers, on gastric tolerance and on treatment adherence (including compliance and persistence).

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women (at least 5 years after natural / surgical menopause).
* Patients on treatment with alendronate 70mg tablets or alendronate 70mg effervescent tablets for 6-8 months and who will be continued to be treated for a minimum of 12 months.
* Available BTMs (s-CTX), biochemistry (calcium, phosphate, 25-OH vit D, PTH, creatinine) and DXA (lumbar spine, total hip and femoral neck) at the initiation of the treatment.
* Ability to sign an informed patient consent

Exclusion Criteria:

* Patients who had received a prior osteoporosis treatment with anti-resorptive drugs (bisphosphonate or denosumab) or teriparatide before starting alendronate 70 mg.
* Any secondary cause of osteoporosis including current treatment with glucocorticoids or aromatase inhibitors, inflammatory disorders, malabsorption
* Metabolic or cancer bone disease
* Contra-indications to bisphosphonates according to product labelling
* Known or suspected allergy to study product(s) or related products
* Inability to sign an informed consent
* Previous participation in this study

Ages: 55 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-menopausal women with osteoporosis, on treatment with Fosamax® or Binosto® for 6-8 months and who will be continued to be treated for a minimum of 12 months, with available BTMs, biochemistry and DXA at the initiation are to be offered participation in the study at the discretion of the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-02-25 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
s-CTX | Change at 6 months, 12 months, 18 months after treatment start
  Decrease in the rate of the bone resorption marker s-CTX

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie TIREFORD, PharmD, Study Director — Labatec Pharma SA
Locations (2):
- Switzerland (2):
  - Endokrinologische Praxis & Labor, Basel, Canton of Basel-City
  - Hôpital Universitaire de Genève, Service des maladies osseuses, Geneva, Canton of Geneva

IPD SHARING:
Plan to Share IPD: No